CLINICAL TRIAL: NCT02761226
Title: Clinical and Radiographic Evaluation of Crestal Bone Loss Around Implant With or Without Platform Switching Design (Randomized Clinical Trial, Split Mouth Design)
Brief Title: Clinical and Radiographic Evaluation of Crestal Bone Loss Around Implant With or Without Platform Switching Design
Acronym: PS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Asma Serag, assisstant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20008
Record Dates: First submitted 2016-04-05; First posted 2016-05-04 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-04

CONDITIONS: Crestal Bone Loss
Keywords: platform switching; dental implant; crestal bone level; implant stability; postoperative complication
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Platform Matched Design) (Experimental): 10 Patients with missing tooth in upper posterior area will receive dental implant (implants with the same abutment diameter)
  Interventions: Procedure: Platform Matched Design (Group A)
- Group B (intervention - Platform Switching Design) (Active Comparator): 10 patients with missing tooth in upper posterior area will receive dental implant (implants with smaller diameter abutment)
  Interventions: Procedure: Platform Switching Design (Group B)

INTERVENTIONS:
Procedure: Platform Matched Design (Group A) — 10 patients with missing upper posterior teeth will receive dental implant with platform matched design (the patients will receive implant 4.2mm with same abutment diameter 4.2mm)
  Other Names: group 1
  Arms: Group A (Platform Matched Design)
Procedure: Platform Switching Design (Group B) — 10 patients with missing upper posterior teeth will receive dental implant with platform switching design(the patients will receive implant 4.2mm with smaller abutment diameter 3.5 mm
  Other Names: group 2
  Arms: Group B (intervention - Platform Switching Design)

SUMMARY:
Implants have become the preferred method of single tooth replacement these days, patients receiving implant treatments not only expect restoration of masticatory function, they also expect that the prostheses will be esthetically pleasing, easy to clean, and permanent. To maintain long-term implant stability, it is important to minimize bone loss around the implant, as well as the soft tissue atrophy that accompanies it.

DETAILED DESCRIPTION:
The peri-implant bone level has been used as one of the criteria to assess the success of dental implants, Platform switching (PLS) for maintaining peri-implant bone levels has gained popularity among implant manufacturers over the last few years. However, the assumption that the inward shifting of the implant- abutment junction may preserve crestal bone was primarily based on serendipitous finding rather than scientific evidence.

It is known that saucerization around an implant occurs following abutment connection using a submerged implant with a butt joint (a two-stage approach), such as the Branemark implant. The nature of saucerization varies according to implant type (one-stage or two-stage) and abutment connection type. they have reported that the factors that are the most likely causes of early crestal bone loss around implants are:

1. The micro-gap,
2. The implant crest module,
3. Occlusal overload, and
4. The biologic width around the dental implant. At the Toronto Conference 1998, the consensus with respect to bone loss around the implant was that bone loss of up to approximately 2 mm during the first year of implant function is acceptable, and at this level the implant is regarded as successful. There have been many reports on studies to ascertain the causes of bone loss around implants and clinical techniques to prevent it. Some reports published in 2005 and 2006 state that the platform switching technique, a technique in which an abutment that is one-size smaller than the implant platform is placed, prevents bone loss around the implant. However, there are only a few reports on the mechanism of action or the extent of bone loss prevention, and as such, it is difficult to say that the effect of PLS has been thoroughly examined. This review article examines the PLS technique and the bone loss preventive effect.

A lot of clinical studies discussed the concept of platform switching was extensively studied histologically and biomechanically. In histomorphometric studies in dogs was no significant difference in the marginal bone level around platform- switched and -matched implants after 28 days of healing. In contrast, other studies reported a significantly less bone loss around platform-switched implants after a loading period of 2 to 6months.

However, there is no consistency among the studies with respect to the study design (e.g. the location and depth of the implant, and controlled/non-controlled), and as such, it is difficult to evaluate all of these studies using the same evaluation method.

The review and meta-analysis show that platform switching may preserve interimplant bone height and soft tissue levels. The degree of marginal bone resorption is inversely related to the extent of the implant- abutment mismatch. But still no general agreement to confirm the validity of this concept, so Further long-term, well-conducted, randomized controlled studies are needed to confirm the validity of this concept.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than18 yrs.
2. Patients with missing teeth in the posterior maxilla (from the 1st premolar to 2nd Molar) bilaterally in need for fixed implant-supported prosthesis.
3. Full mouth plaque score and full mouth bleeding score ˂25 %
4. Patients with adequate bone quality and quantity at the implant site
5. Patients with systematic healthy.
6. Non-smokers or those smoking ˂10 cigarettes/day
7. Patients who were cooperative, motivated, and hygiene conscious and willing to return for multiple follow-up appointments (up to 9 months after prosthetic loading).

Exclusion Criteria:

I) General:-

1. Patients with any systemic condition that may contraindicate implant therapy.
2. Patients with a history of Bisphosphonate therapy
3. Pregnant and lactating patients
4. Alcohol and drug abuse
5. Parafunctional habits that produce overload on the implant such as bruxism and clenching.

II) Local:-

1. Local inflammation or infection at implant site.
2. Untreated periodontitis
3. Local irradiation therapy
4. History of implant failure as well as unhealed extraction socket
5. Inadequate keratinized gingiva or thin gingival biotype.
6. Inadequate bone height or width.
7. Insufficient vertical inter-arch space, upon centric occlusion, to accommodate the available restorative components.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
crestal bone loss | 9 months
  assessment crestal bone loss after 9 months after crown placement

SECONDARY OUTCOMES:
implant stability | 9 months
  assessment implant placement by periotest at abutment instillation and after 9 month of crown placement

IPD SHARING:
Plan to Share IPD: Undecided